CLINICAL TRIAL: NCT00073541
Title: An Open-Label Phase II Study in Subjects With Recurrent EGFR-Positive Ovarian Cancer to Investigate the Safety and Efficacy of EMD 72000 Administered as a Single Agent
Brief Title: A Study of the Safety and Effects of EMD 72000 in Subjects With Recurrent Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: EMD Serono (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: EMD 72000-030
Record Dates: First submitted 2003-11-24; First posted 2003-11-26 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Ovarian Cancer
Keywords: EGFR; HER-1; monoclonal antibody; targeted therapy
MeSH Terms: conditions — Ovarian Neoplasms | interventions — matuzumab

INTERVENTIONS:
Drug: EMD 72000

SUMMARY:
EMD 72000 is an experimental, biological drug. Studies in animals indicate that EMD 72000 blocks a factor found on the surface of many cancer cells. The factor is called epidermal growth factor receptor or EGFR. One type of cancer which frequently contains EGFR is ovarian cancer. This study will test the safety and effects of EMD 72000 in subjects with EGFR-positive recurrent ovarian cancer following standard treatment that has failed.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent ovarian cancer (including primary peritoneal cancer) following treatment (e.g., doxorubicin HCL liposome, topotecan, etc.) for primary or secondary platinum-refractory disease
* Immunohistochemical evidence of tumor EGFR (HER-1) expression
* At least one measurable lesion according to the WHO criteria
* Life expectancy ≥ 12 weeks
* ECOG performance status 0-1

Exclusion Criteria:

* History of prior MAb therapy
* History of prior treatment with an EGFR (HER-1) directed therapy
* Known brain metastases
* Presence of a ≥ Grade 2 pre-existing skin disorder (alopecia is permitted)
* Known intercurrent infections or immunosuppression
* Actively infected with, or chronic carriers of HBV
* Evidence of HCV disease
* Previous diagnosis of autoimmune disease
* Known hypersensitivity to the administered drugs or any of their components
* Receipt of chemotherapy, radiation therapy, or another investigational drug within 30 days of enrollment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2003-04; Primary Completion 2004-03 (Actual); Study Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Baltimore, Maryland
  - Boston, Massachusetts
  - New York, New York
  - Charlotte, North Carolina
  - Nashville, Tennessee

REFERENCES:
- [Result] Seiden MV, Burris HA, Matulonis U, Hall JB, Armstrong DK, Speyer J, Weber JD, Muggia F. A phase II trial of EMD72000 (matuzumab), a humanized anti-EGFR monoclonal antibody, in patients with platinum-resistant ovarian and primary peritoneal malignancies. Gynecol Oncol. 2007 Mar;104(3):727-31. doi: 10.1016/j.ygyno.2006.10.019. Epub 2006 Nov 28. PMID 17126894